CLINICAL TRIAL: NCT06220838
Title: A Phase Ⅰ Study to Evaluate the Safety/Tolerability, Pharmacokinetics, and Efficacy of SC-101 in Subjects With Advanced or Metastatic Solid Tumors That Express Nectin-4
Brief Title: Study SC-101 in Subjects With Advanced Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin ConjuStar Biologics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-101-101
Record Dates: First submitted 2024-01-12; First posted 2024-01-24 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SC-101 (Experimental)
  Interventions: Drug: SC-101

INTERVENTIONS:
Drug: SC-101 — All subjects will receive a single intravenous (IV) infusion of SC-101 once weekly.

SUMMARY:
This study will evaluate the safety, pharmacokinetics, and anti-cancer efficacy of SC-101 in subjects with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
This study is the first-in-human (FIH), multi-center, open-label trial of SC-101, including the dose escalation and expansion phases.

The dose escalation study is primarily designed to assess the safety and tolerability of SC-101 and to determine the recommended dose(s) for the dose expansion study. The dose expansion study is designed with the primary objective of evaluating the clinical activity of SC-101 in patients with metastatic urothelial carcinoma or other solid tumors that express Nectin-4.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily agree to participate in the study and sign the Informed Consent Form (ICF).
2. 18 to 80 years of age at the time of signature of the ICF, without gender limitation.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Life expectancy of ≥ 3 months as assessed by the investigator.
5. Women and men of childbearing potential must be advised and agree to practice effective methods of contraception during the study.
6. Understand study requirements, and willing and able to comply with arrangements of study and follow-up procedures.
7. Adequate Bone Marrow Reserve and Organ Functions.
8. Subjects must have measurable disease according to RECIST (version 1.1).
9. Histologically or cytologically confirmed advanced malignant solid tumors.
10. For non-urothelial carcinoma patients enrolled in the dose expansion study: Subjects must have a positive expression of Nectin-4 in their tumor samples as confirmed by the central laboratory.
11. Subjects are willing to follow study procedures.

Exclusion Criteria:

1. History of other malignancy(ies) within 3 years before signing the ICF, except for non-melanoma skin cancer, cervical carcinoma in situ, or other malignant tumors that are considered to have been cured.
2. Any anticancer therapy, including any investigational drug, within 2 weeks before the first dose of the study drug.
3. Uncontrolled central nervous system metastases.
4. Prior treatment with Nectin-4-targeting anti-cancer therapy.
5. Preexisting treatment-related toxicity Grade ≥ 2 (except alopecia).
6. Preexisting Grade ≥ 2 (as per CTCAE v5.0) sensory or motor neuropathy.
7. Major surgery within 4 weeks prior to the first dose of the study drug.
8. History of interstitial lung disease (ILD), preexisting ILD, or the suspected ILD that cannot be ruled out by imaging examination at screening.
9. Preexisting active keratitis or corneal ulcerations.
10. Preexisting serious dermatological diseases, or having experienced serious skin toxicities during the prior anti-cancer treatment (e.g., Stevens-Johnson syndrome, toxic Epidermal Necrolysis, etc.).
11. Currently receiving systemic antimicrobial treatment for active infection (viral, bacterial, or fungal) at the time of first dose of study drug, or fever within 14 days prior to the first dose of the study drug.
12. History of uncontrolled diabetes mellitus.
13. History of thromboembolic events and bleeding disorders ≤ 6 months (e.g.,deep vein thrombosis (DVT) or pulmonary embolism ( PE)) prior to the first dose of the study drug.
14. Positive results of virus serology tests.
15. History of serious cardiovascular and cerebrovascular diseases, including but not limited to:

    1. Serious cardiac arrhythmias or conduction abnormalities, such as ventricular arrhythmia require treatment, and grade 2 or 3 atrioventricular block.
    2. QTc prolongation to >450 milliseconds (ms) in males and >470 ms in females based on ECG.
    3. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or transient ischemic attack (TIA) within 6 months prior to the first dose of the study drug.
    4. New myocardial infarction or unstable angina within 6 months before the first dose of the study drug.
    5. Uncontrolled hypertension.
16. Require ongoing therapy with a medication that is a strong inhibitor or inducer of the cytochrome P450 3A4 (CYP3A4) enzymes.
17. Known sensitivity to any of the ingredients of the investigational product.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (dose escalation phase) | Up to 30 days after the last dose of study drug
Objective response rate (dose expansion phase) | Every 8 weeks (± 7 days)
  Defined as the percentage of subjects who experience a best response of either complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of SC-101 and monomethyl auristatin E (MMAE) when given as monotherapy | From Cycle 1 Day 1 through end of treatment (EOT)
  Plasma concentrations of SC-101 and MMAE from all participants taking SC-101 alone
Minimum plasma concentration (Cmin) of SC-101 and monomethyl auristatin E (MMAE) when given as monotherapy | From Cycle 1 Day 1 through end of treatment (EOT)
  Plasma concentrations of SC-101 and MMAE from all participants taking SC-101 alone
Area under the plasma concentration-time curve (AUC) of SC-101 and monomethyl auristatin E (MMAE) when given as monotherapy | From Cycle 1 Day 1 through end of treatment (EOT)
  Plasma concentrations of SC-101 and MMAE from all participants taking SC-101 alone
Elimination half-life (t1/2) of SC-101 and monomethyl auristatin E (MMAE) when given as monotherapy | From Cycle 1 Day 1 through end of treatment (EOT)
  Plasma concentrations of SC-101 and MMAE from all participants taking SC-101 alone
Number of participants positive for anti-drug antibodies (ADA) | From Cycle 1 Day 1 through end of treatment (EOT)
  Number of participants positive for anti-drug antibodies (ADA) from all participants receiving SC-101 monotherapy
Duration of Response (DoR) | Every 8 weeks (± 7 days)
  Defined as the time from first assessment of partial response (PR) or complete response (CR) until disease progression.
Disease Control Rate (DCR) | Every 8 weeks (± 7 days)
  Defined as the percentage of subjects who experience a best response of either complete response (CR), partial response (PR) or stable disease (SD).

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No